CLINICAL TRIAL: NCT04938973
Title: Near-Infrared Fluorescence-Guided Robotic-Assisted Minimally Invasive Esophagectomy Using Indocyanine Green Dye Versus Open Transthoracic Esophagectomy: A Randomized Controlled Feasibility Trial
Brief Title: NIF-Guided RAMIE Using ICG Versus OTE Feasibility RCT
Acronym: RAMIE vs OTE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was closed due to adverse events because the adverse event rate was not lower than the adverse event rate in traditional open esophagectomy.
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Wael Hanna, Associate Professor, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJHH_RAMIE_vs_OTE_Feasibility
Record Dates: First submitted 2021-06-08; First posted 2021-06-25 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NIF-Guided RAMIE using ICG Dye (Experimental Arm) (Experimental): The patient will undergo NIF-guided RAMIE using ICG dye using the standard Ivor-Lewis approach. This will be a two-stage operation involving a first stage through a 5-port robotic approach through the abdomen to achieve a proximal gastrectomy and D2 nodal dissection. A feeding jejunostomy would not be inserted, as per the enhanced recovery pathway for esophagectomy. In addition, the vascularization of the conduit can be confirmed using the near-infrared camera of the robot with the ICG dye. The second stage of the operation will involve a 4-port robotic approach through the right chest to achieve thoracic nodal dissection, esophagectomy, and a hand-sewn anastomosis between the residual esophagus and the gastric conduit at the level of the azygous vein. During this second stage of the operation, NIF with ICG dye will be used to visualize the vascular supply of the gastric conduit, and assess the gastric conduit for any perfusions to potentially reduce anastomotic leaks.
  Interventions: Procedure: Robotic Assisted Minimally Invasive Esophagectomy (RAMIE); Device: Robotic Assisted Minimally Invasive Esophagectomy (RAMIE)
- Open Transthoracic Esophagectomy (OTE) (Active Comparator): The patient will undergo OTE using the standard Ivor-Lewis approach. This is a two-stage operation involving a first stage through laparotomy, proximal gastrectomy, D2 nodal dissection, and insertion of feeding jejunostomy. The second stage of the operation will involve a right thoracotomy, thoracic nodal dissection, esophagectomy, and a stapled anastomosis between the residual esophagus and the gastric conduit at the level of the azygous vein.
  Interventions: Procedure: Open Transthoracic Esophagectomy (OTE)

INTERVENTIONS:
Procedure: Robotic Assisted Minimally Invasive Esophagectomy (RAMIE) — Robotic Assisted Minimally Invasive Esophagectomy (RAMIE) will be performed using the Da Vinci Robotic Surgical Platform.
  Arms: NIF-Guided RAMIE using ICG Dye (Experimental Arm)
Procedure: Open Transthoracic Esophagectomy (OTE) — Open Transthoracic Esophagectomy (OTE) is the current standard of care.
  Arms: Open Transthoracic Esophagectomy (OTE)
Device: Robotic Assisted Minimally Invasive Esophagectomy (RAMIE) — Robotic Assisted Minimally Invasive Esophagectomy (RAMIE) will be performed using the Da Vinci Robotic Surgical Platform.
  Arms: NIF-Guided RAMIE using ICG Dye (Experimental Arm)

SUMMARY:
In Canada, the incidence of esophageal cancer has been increasing over time, while surgical standards for esophageal resections have remained unchanged. Currently, the standard of surgical care for this cancer is Open Transthoracic Esophagectomy (OTE), a highly morbid operation that is associated with a complication rate of 60-80%, and a recovery period of many months. While Minimally Invasive Esophagectomy (MIE) has been developed it has not been adopted because it is highly complex, technically demanding, and has a longer operative time than OTE. With the advent of robotic platforms, Robotic Assisted Minimally Invasive Esophagectomy (RAMIE) has recently emerged as a novel minimally invasive alternative to OTE. RAMIE utilizes the DaVinci Xi robotic surgical platform which offers superior dexterity, 3D-vision, and wristed surgical equipment. To date, case reports and small case series have demonstrated the safety of RAMIE, however it has not been performed yet in Canada, and there has been no randomized trial that has compared RAMIE to OTE. This study proposes to build the infrastructure for introducing RAMIE to Canada, while laying the foundations for a future randomized controlled trial which will compare it to OTE.

DETAILED DESCRIPTION:
In Canada, the incidence of esophageal cancer has been increasing over time. The treatment of patients with cancer of the esophagus is multi-modal, with surgery being the cornerstone of most treatment regimens. Operative treatment is usually performed through Open Transthoracic Esophagectomy (OTE), a highly morbid procedure that is associated with a complication rate of 60-80%, and a recovery period of many months. This standard is being challenged by a growing body of evidence demonstrating that a minimally invasive approach can reduce post-operative morbidity and improve quality-of-life, while still offering an adequate oncological outcome. The minimally invasive alternative to OTE is Minimally Invasive Esophagectomy (MIE). Although MIE has been shown to reduce the morbidity associated with esophagectomy, it has not been widely adopted. This failure of adoption is due to the high complexity of MIE; it is an exceedingly difficult operation, is associated with a very steep learning curve, and can take 8-10 hours to complete. As a result, less than 10% of esophageal cancer programs in Canada have adopted MIE, and there remains a need for a minimally invasive alternative to OTE. Robotic Assisted Minimally Invasive Esophagectomy (RAMIE) has recently emerged as a minimally invasive alternative to OTE. RAMIE utilizes the DaVinci Xi robotic surgical platform which offers superior dexterity, 3D-vision, 7-degrees of freedom for range of motion, and near-infrared imaging for detection of blood vessels. As a result, RAMIE has succeeded where MIE has failed, and has been widely taken up in Europe and the United States.

To date, near-infrared fluorescence (NIF)-guided RAMIE using indocyanine green (ICG) dye has not been performed in Canada, and there has been no randomized trial that has compared NIF-guided RAMIE using ICG dye to OTE. In this study, we propose to build the infrastructure for introducing NIF-guided RAMIE using ICG dye to Canada, while laying the foundations for a future randomized controlled trial (RCT) which will compare it to OTE. This study is a Phase I, single center, prospective feasibility randomized controlled trial with two phases: Phase A: Learning Curve of NIF-guided RAMIE using ICG dye; and Phase B: A Randomized Controlled Feasibility Trial. In Phase A, 40 patients will be enrolled, and they will all undergo NIF-guided RAMIE using ICG dye. Evidence shows that a surgeon experienced in MIE requires experience of 40 cases to gain proficiency of RAMIE. In Phase B, 54 patients will be enrolled, and they will be randomized to either NIF-guided RAMIE using ICG dye, or OTE.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Clinical Stage I, II, or III esophageal cancer, who are candidates for surgery after discussion in multidisciplinary tumor board.
* Candidates for minimally invasive surgery as determined by the operating surgeon.

Exclusion Criteria:

* Hypersensitivity or allergy to ICG, sodium iodide, or iodine
* Women who are currently pregnant or are breastfeeding; or women of childbearing potential who are not currently taking adequate birth control
* Clinical Stage IV esophageal cancer.
* Not a candidate for minimally invasive surgery as determined by the operating surgeon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
The feasibility of a large-scale RCT, as measured by the number of patients willing to participate in the study. | 3-Weeks Postoperative
  A recruitment rate ≥70%, whereby participants partake in the study until first post-operative follow-up, would be considered acceptable.

SECONDARY OUTCOMES:
Safety of the Operation, based on rates of perioperative complications | 12-Weeks Postoperative
  The safety of the operation based on rates of perioperative complications within 90-days of surgery, as defined by the Ottawa Thoracic Morbidity and Mortality Classification System (TMNM).
Patient-Reported Health-Related Quality of Life - Pain Level | Baseline, Postoperative Day 1, 3-Weeks Postoperative, 12-Weeks Postoperative
  The Stanford Pain Scale will be administered to patients to assess pain (0 = no pain, 10 = worst pain)
Patient-Reported Health-Related Quality of Life - Quality of Life | Baseline, Postoperative Day 1, 3-Weeks Postoperative, 12-Weeks Postoperative
  EQ-5D-5L will be administered to patients to assess pain and quality of life. 5 items + overall health rating (0-100; 0 worst health imaginable, 100 best health imaginable)
Patient-Reported Health-Related Quality of Life - Reintegration into Normal Living | Baseline, Postoperative Day 1, 3-Weeks Postoperative, 12-Weeks Postoperative
  Reintegration to Normal Living Index will be administered to patients to assess quality of life. 11 items, each item scored from 1-10 (1 = no reintegration, 10 = complete reintegration)
Conversion from RAMIE to OTE | During Surgery
  Rate of conversions from RAMIE to OTE
Length of Stay (LOS) | From Date of Admission to Date of Discharge, assessed up to 12-Weeks Postoperative
  Length of hospital stay will be measured between the date of admission and date of discharge.
Length of Operation | During Surgery
  Operative time will be measured by collecting the procedure start and procedure end time

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No